CLINICAL TRIAL: NCT04346394
Title: The Role of the Noradrenergic System in the Nonmotor Symptoms of Parkinson's Disease: Orthostatic Hypotension and Other Nonmotor Symptoms
Brief Title: The Role of the Noradrenergic System in the Nonmotor Symptoms of Parkinson's Disease
Acronym: NAinPD
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: COVID-19
Sponsor: Nathaniel M. Robbins (Other)
Responsible Party: Sponsor-Investigator, Nathaniel M. Robbins, Physician, Assistant Professor of Neurology, Dartmouth-Hitchcock Medical Center
Organization: Dartmouth-Hitchcock Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: D19090
Record Dates: First submitted 2020-03-10; First posted 2020-04-15 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Parkinson Disease
Keywords: Parkinson's; Orthostatic Hypotension; Yohimbine
MeSH Terms: conditions — Parkinson Disease; Hypotension, Orthostatic | interventions — Yohimbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Yohimbine (Experimental): The first visit in the study has no interventional drug. Yohimbine (5mg) is administered orally during visit two, during a head up tilt test, to manipulate the noradrenergic system to determine the association between OH and NP symptoms in those with PD. Yohimbine is not administered as a treatment in this study, but as a pharmacologic tool to study the adrenergic system.
  Interventions: Drug: Yohimbine HCl

INTERVENTIONS:
Drug: Yohimbine HCl — Yohimbine hydrochloride will be used to manipulate the noradrenergic system during some of the assessments. By measuring the amounts of hormones the body produces before and after yohimbine hydrochloride administration, researchers can assess how well the noradrenergic system is functioning
  Other Names: Yohimbine hydrochloride, yohimbine

SUMMARY:
The goal of this clinical trial is to learn about the role of noradrenergic system in the non-motor symptoms of Parkinson's disease. The main objectives it aims to answer are:

1. To explore the association between orthostatic hypertension which is low blood pressure that occurs after going from lying to standing, and several neuropsychiatric and neurocognitive nonmotor features of Parkinson's disease (PD), such as feeling tired or disinterested and depression.
2. To explore the association between central noradrenergic dysfunction, orthostatic hypertension, and nonmotor symptoms of PD by measuring hormonal response to head up tilt-table testing before and after administration of yohimbine.
3. To explore the association between central noradrenergic dysfunction, orthostatic hypertension, and nonmotor symptoms of PD by measuring participants pupils before and after administration of yohimbine

Participants will be asked to come onsite for two study visits.

Visit one will consist of:

* Discussing and signing the Informed Consent Form
* Discussing Medical History and Current Medications
* Collecting Blood samples
* Measuring heart rate and blood pressure
* Mental health screening and neurocognitive questionnaires
* Pupil test
* Test to feel vibrations

Visit two will consist of :

* Mental Health questionnaire
* IV Placement
* Blood Draws
* Administration of Yohimbine hydrochloride
* Head up tilt table
* Measuring heart rate and blood pressure
* Answering questions about anxiety, mood, and fatigue using a scale
* Pupil tests

Visit three will be a follow-up call from the Nurse Coordinator to discuss any adverse events.

DETAILED DESCRIPTION:
This is a cross-sectional pilot study comparing 10 PD patients with Orthostatic hypertension (OH) to 10 PD patients without OH. OH is defined as a drop in blood pressure within 5 minutes of standing (measured at 1, 2, and 5 minutes). The study will include two clinical visits and a follow-up phone call 24-72 hours after the 2nd visit. Visits will last approximately 4-5 hours each. During visit two the participant will be given a 5 mg tablet of Yohimbine hydrochloride. Yohimbine hydrochloride will be administered orally during Visit 2 in order to manipulate the noradrenergic system to determine the association between OH and neuropsychiatric symptoms in those with PD. Yohimbine is not administered as a treatment in this study, but as a tool to study the noradrenergic system during some of the assessments. This will be done by measuring the amounts of hormones in the participants body produces before and after yohimbine hydrochloride administration. Yohimbine hydrochloride is not approved by the FDA for this use.

On the morning of Visit 1, the participant will be asked to not take their medications that contains dopamine, such as levodopa/carbidopa, as well as other medications that would interfere with testing. The study doctor will determine which medications need to be held for this visit. The participant will be asked to bring one dose of these medications to take during the visit, instead of at the normal time in the morning. During visit one eligibility criteria will be discussed and if participants meet the inclusion exclusion criteria the Informed Consent will be signed and Visit 1 procedures will follow.

Visit 2 will occur no more than 30 days after visit 1. Subjects will be asked to not eat, and not take morning medications containing dopamine or norepinephrine (such as levodopa/carbidopa), or any other medications that interfere with testing. The neurologist will determine which medications need to be held for this visit. An IV will be placed as per Head Up Tilt procedure. Head Up Tilt testing will be conducted twice, once prior to and once after yohimbine administration. The participant will complete a scale that measures anxiety, mood, and fatigue prior to and after yohimbine administration. Pupil testing will also be evaluated prior to yohimbine administration and after yohimbine administration. Blood will be drawn twice prior to yohimbine administration and twice after yohimbine administration. One draw will be in a lying down position, and the other will be during the head up tilt.

A follow up study phone call will be made by the study nurse coordinator 24-72 hours after study visit 2. Any adverse events which may have occurred since the study visit will be captured on the participants adverse event log.

ELIGIBILITY:
Inclusion Criteria:

1. Participant able to provide informed consent
2. Diagnosis of Parkinson's disease confirmed by a DH neurologist according to Movement Disorder Society criteria, with the exception that "Red flag" 5a will not be used (severe autonomic failure within five years of disease onset).
3. All subjects must have CMP and CBC drawn within 6 months of study visit 1, with results in the normal range or with abnormal results not considered to be clinically significant in the investigator's opinion.
4. Female patients must be post-menopausal (at least one year) or not planning to get pregnant and have negative pregnancy test.

Exclusion Criteria:

1. Diagnosis or previous history of diabetes of any kind
2. Known autonomic neuropathy unrelated to PD
3. History of or current cardiac, liver or renal disease that, in the opinion of the investigator, may put the patient at risk because of participation in the study
4. Known condition that in the investigator's opinion would be a contraindication to HUT testing or yohimbine challenge (e.g. decompensated cardiac disease, severe positional vertigo; severe anxiety, known panic disorder69)
5. Current use of catecholaminergic medications (e.g. stimulants, droxidopa, midodrine) that cannot be held for at least three half-lives
6. Inability to hold PD medications for at least 12 hours
7. History of major depressive or bipolar disorder preceding the diagnosis of PD,69 or diagnosis or previous history of psychiatric illness that in the investigator's opinion would affect the subject's ability to successfully participate in the study.
8. Any history (other than PD) that could significantly and adversely affect neurocognitive function, such as history of traumatic brain injury (head injury with loss of consciousness > 1 hour), known dementia unrelated to Parkinson's or related diseases; developmental delay, multiple sclerosis or epilepsy with cognitive impairment, intellectual deficit, diagnosed and untreated sleep apnea; untreated syphilis; HIV with HAND; or other conditions that, based on the investigators opinion, could interfere with neurocognitive evaluation.
9. Known ophthalmologic disease such as untreated cataract, glaucoma, optic neuritis, orbital trauma, or other neuroretinal disease that might impact pupillary function
10. Severe illness within 30 days prior to enrollment.
11. Use of opiate, procholinergic, or other medications influencing pupillary function that cannot be held for three half-lives
12. In the Investigator's opinion, subject would be unable to successfully participate in the study for any reason.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-05-11 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Difference in fatigue (measured with the self-reported Fatigue Severity Scale) in patients with Parkinson's disease with and without orthostatic hypotension (PD+OH v PD-OH) | All measurements for this study will be obtained during one of the two study visits that each subject will undergo. These two visits will be completed within 6 months of subject enrollment
  The Fatigue Severity Scale (FSS) measures average fatigue experienced over the previous week. The FSS questionnaire contains nine statements that rate the severity of fatigue symptoms. A low value indicates strong disagreement with the statement, a high value indicates strong agreement. A total score of 36 or more suggests presence of fatigue.

SECONDARY OUTCOMES:
Difference in apathy (measured with the self-reported Apathy Evaluation Scale) in patients with Parkinson's disease with and without orthostatic hypotension (PD+OH v PD-OH) | All measurements for this study will be obtained during one of the two study visits that each subject will undergo. These two visits will be completed within 6 months of subject enrollment
  Apathy Evaluation Scale (AES) measures apathy over the previous month. The AES questionnaire contains 18 statements that each rAll measurements for this study will be obtained during one of the two study visits that each subject will undergo. These two visits will be completed within 6 months of subject enrollment ate the severity of apathy on a scale from 1 to 4. A total score ranges from 18 to 72, with higher scores indicating more apathy.
Difference in self-reported depression (measured with the Geriatric Depression Scale - short form) in patients with Parkinson's disease with and without orthostatic hypotension (PD+OH v PD-OH) | All measurements for this study will be obtained during one of the two study visits that each subject will undergo. These two visits will be completed within 6 months of subject enrollment
  The Geriatric Depression Scale - short form measures depression over the previous week. This questionnaire contains 15 questions that are answered by either indicating "Yes" or "No" to the questions. The total score ranges from 0 to 15, with higher scores indicating more depression.
Difference in self-reported anxiety (measured with the Geriatric Anxiety Inventory) in patients with Parkinson's disease with and without orthostatic hypotension (PD+OH v PD-OH) | All measurements for this study will be obtained during one of the two study visits that each subject will undergo. These two visits will be completed within 6 months of subject enrollment
  The Geriatric Anxiety Inventory measures anxiety over the previous week. This questionnaire contains 20 questions that are answered by indicating either "Yes" or "No" to the questions. The total score ranges from 0 to 20, with higher scores indicating more anxiety.
Difference in neurocognition (measured with average composite z-score on a neurocognitive battery) in patients with Parkinson's disease with and without orthostatic hypotension (PD+OH v PD-OH) | All measurements for this study will be obtained during one of the two study visits that each subject will undergo. These two visits will be completed within 6 months of subject enrollment
  Neurocognition will be measured with the following battery, adjusting for age, gender, education level, and premorbid functioning. Digit Span subtest from the Wechsler Adult Intelligence Scale - IV; Symbol Digit Modalities Test; Trail Making Test; California Verbal Learning Test - II; Rey Complex Figure Test; DKEFS Color-Word Interference Test; Phonemic and Semantic Verbal Fluency; Behavior Rating Inventory of Executive Function - Adult Outcome. An average composite z-score will calculated and compared between groups.
Difference in informant-reported anxiety (measured by an informant-reported Neuropsychiatric Inventory Questionnaire) in patients with Parkinson's disease with and without orthostatic hypotension (PD+OH v PD-OH). | All measurements for this study will be obtained during one of the two study visits that each subject will undergo. These two visits will be completed within 6 months of subject enrollment
  The NPI-Q measures 12 psychiatric symptoms, and each symptom (ie anxiety) is scored as absent or present.
Difference in informant-reported apathy (measured by an informant-reported Neuropsychiatric Inventory Questionnaire) in patients with Parkinson's disease with and without orthostatic hypotension (PD+OH v PD-OH) | All measurements for this study will be obtained during one of the two study visits that each subject will undergo. These two visits will be completed within 6 months of subject enrollment
  The NPI-Q measures 12 psychiatric symptoms, and each symptom (ie apathy) is scored as absent or present.
Difference in informant-reported depression (measured by an informant-reported Neuropsychiatric Inventory Questionnaire) in patients with Parkinson's disease with and without orthostatic hypotension (PD+OH v PD-OH). | All measurements for this study will be obtained during one of the two study visits that each subject will undergo. These two visits will be completed within 6 months of subject enrollment
  The NPI-Q measures 12 psychiatric symptoms, and each symptom (ie depression) is scored as absent or present
Change in serum catecholamine levels (supine and orthostatic) before and after yohimbine administration | Baseline (supine position), after 5 minutes of head-up tilt, 60 minutes after yohimbine administration (supine position), and 5 minutes after that with repeat head-up tilt.
  Change in serum catecholamine levels will be measured from blood samples collected from participants upon lying face up and 5 minutes after head-up tilt, before and after yohimbine administration
Change in serum desmopressin levels (supine and orthostatic) before and after yohimbine administration | Baseline (supine), after 15 minutes of head-up tilt, 60 minutes after yohimbine administration (supine position) and 15 minutes after that with repeat head-up tilt
  Change in serum desmopressin levels 15 minutes after head-up tilt before and after yohimbine administration

OTHER OUTCOMES:
Between group (Parkinson patients with and without orthostatic hypotension (PD+OH v PD-OH) change in self-reported anxiety before and after yohimbine administration | Baseline and 45 minutes after yohimbine administration
  Change in self-reported anxiety levels before and after yohimbine administration measured with an 11-point visual analogue scale (0-10), where a higher score indicate more anxiety and fatigue
Between group (Parkinson patients with and without orthostatic hypotension (PD+OH v PD-OH) change in self-reported mood before and after yohimbine administration | Baseline and 45 minutes after yohimbine administration
  Change in self-reported mood before and after yohimbine administration measured with an 11-point visual analogue scale (0-10), where a higher score indicate more anxiety and fatigue
Between group (Parkinson patients with and without orthostatic hypotension (PD+OH v PD-OH) change in self-reported fatigue before and after yohimbine administration | Baseline and 45 minutes after yohimbine administration
  Change in self-reported fatigue levels before and after yohimbine administration measured with an 11-point visual analogue scale (0-10), where a higher score indicate more anxiety and fatigue
Between group (PD+OH v PD-OH) change in diastolic blood pressure before and after yohimbine | Baseline (after resting 30 minutes supine) and 45 minutes after yohimbine administration
  Change in diastolic blood pressure (measured in mmHg, supine after 30 min rest) before and after yohimbine administration in Parkinson's patient with and without orthostatic hypotension
Between group (PD+OH v PD-OH) change in time until pupillary redilation before and after yohimbine | Baseline (after resting 30 minutes supine) and 45 minutes after yohimbine administration
  Change in time until pupillary redilation (measure in seconds after brief light stimulus using a NeuroOptics pupilometer) before and 45 minutes after yohimbine administration
Between group (PD+OH v PD-OH) difference in change in time to recovery of BP after 60 degree head-up tilt before and after yohimbine administration | Baseline tilt test before yohimbine and second tilt 60 minutes after yohimbine administration
  Change in time to recovery of systolic blood pressure (measured in seconds back to baseline) after 60 degree head-up tilt before and after yohimbine administration

CONTACTS AND LOCATIONS:
Overall Officials: Nathaniel M Robbins, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock, Lebanon, New Hampshire, United States

DOCUMENTS (1):
  • Study Protocol (2019-11-14): https://cdn.clinicaltrials.gov/large-docs/94/NCT04346394/Prot_000.pdf